CLINICAL TRIAL: NCT06224062
Title: Comparison of SARS-CoV-2, AdenoVIRus and Rhinovirus Infection of the Respiratory Epithelium in CHILdren vs. the eLDerly
Brief Title: Virus and Bronchial Epithelium in Children and the Elderly
Acronym: VIRCHILLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2021/43
Record Dates: First submitted 2023-12-22; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-12

CONDITIONS: SARS-CoV-2
Keywords: Adenovirus; SARS-COV-2; Rhinovirus; Children; Elderly
MeSH Terms: conditions — Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- children (Experimental): reconstituted fully functional respiratory epithelium obtained from children (0 -18 years old)
  Interventions: Biological: SARS-CoV-2; Biological: Adenovirus (AdV); Biological: Rhinovirus; Biological: No Intervention
- adults (Experimental): reconstituted fully functional respiratory epithelium obtained from adults (18 to 60 years old)
  Interventions: Biological: SARS-CoV-2; Biological: Adenovirus (AdV); Biological: Rhinovirus; Biological: No Intervention
- elderly (Experimental): reconstituted fully functional respiratory epithelium obtained from adults (over 60 years old)
  Interventions: Biological: SARS-CoV-2; Biological: Adenovirus (AdV); Biological: Rhinovirus; Biological: No Intervention

INTERVENTIONS:
Biological: SARS-CoV-2 — Circulating strains of SARS-CoV-2 (including variants of concern) were already collected, cultured and purified. The Wuhan reference strain will be used in the VIRCHILLD study to infect cells.
Biological: Adenovirus (AdV) — Infection with C-type viruses (e.g. HAd-C5) using bronchial epithelium from adult donors
Biological: Rhinovirus — RV is a member of the picornaviridae family; small non-enveloped viruses with a single strand positive RNA genome protected by an icosahedral capsid. They are divided in more than 160 serotypes classed in subtype A, B and C. RV-A and RV-C infections will be used in the VIRCHILLD study
Biological: No Intervention — no infection

SUMMARY:
The objective of the VIRCHILLD project is to identify age-related modifications of the bronchial epithelium physiology that account for differences in the response and susceptibility to respiratory viruses. Epidemiology and cell-based data show that respiratory virus infections differentially affect children, adults or the elderly populations.

The current worldwide pandemic of SARS-CoV-2 clearly highlighted this notion with a large part of the deaths occurring in the elderly population and very few deaths amongst children. This may be linked to a decreased transmission and/or viral load with SARS-CoV-2 in children compared to adults and elderly. Less in the public eye is the observation that other major respiratory virus targeting the bronchial epithelium (BE) such as rhinovirus (RV) and adenovirus (AdV) cause important clinical feature in children and have a much lower incidence in adults and the elderly populations, which is the opposite to the situation with SARS-CoV-2. Based on this remarkable discrepancy between respiratory viruses the investigators hypothesize that intrinsic age-controlled properties of the respiratory epithelium under resting physiological conditions determine virus susceptibility and virus propagation.

DETAILED DESCRIPTION:
The objective of the VIRCHILLD project is to identify age-related modifications of the bronchial epithelium physiology able to explain differences in the response to respiratory viruses. Several epidemiological and cell-based data have demonstrated that respiratory virus infections differentially affect children, adults or the elderly populations. Perhaps, this difference has been put most notably into the spotlight by the current worldwide pandemic of SARS-CoV-2 with a large part of the deaths occurring in the elderly population whereas very few deaths amongst children have been recorded. According to some studies, this could be linked to a decreased transmission and/or viral load with SARS-CoV-2 in children compared to adults and elderly. What is less in the public eye is the observation that other major respiratory virus targeting the bronchial epithelium such as rhinovirus and adenovirus cause important clinical feature in children and have a much lower incidence in adults and the elderly populations, which is the opposite to the situation with SARS-CoV-2. Based on this remarkable discrepancy between respiratory viruses the investigators hypothesize that intrinsic age-controlled properties of the respiratory epithelium under resting physiological conditions determines virus susceptibility and virus propagation. Such hypothesis is supported by the literature and our own strong preliminary data. A highly complementing consortium composed of experts in lung physiology, pulmonary transcriptomic, respiratory viruses and ultrastructure analysis will address the question. The investigators will use three major respiratory pathogens (AdV, RV and SARS-CoV-2) to infect reconstituted fully functional respiratory epithelium obtained from children, adults and elderly and study parameters of virus infection and epithelial response. This project should highlight specific therapeutic targets against respiratory viruses with a high prevalence in children such as rhinovirus and adenoviruses to increase the therapeutic arsenal of clinician against those infections.

ELIGIBILITY:
Inclusion Criteria:

For pediatric patients requiring research-specific bronchial brushing:

* Child under 18 years old,
* Requiring bronchoscopy as part of routine care
* Having informed and signed consent from the holders of parental authority

For pediatric patients whose bronchial brushing will be carried out as part of their care and for those whose surgical waste will be collected for research:

* Child under 18 years old,
* Requiring as part of routine care bronchoscopy and brushing or bronchial fibroscopy under general anesthesia or surgical resection/lobectomy
* Having expressed their non-opposition to their child's participation in research

For adult patients:

* Man or woman
* Aged 18 or over
* Requiring as part of the care, thoracic surgery such as lobectomy, pneumonectomy or lung transplantation in the Thoracic Surgery Department of Haut Lévêque du Chu Hospital in Bordeaux or inclusion in the TUBE study, described below.
* having received an information note and not having objected to their participation in the research

Exclusion Criteria:

* No affiliation or non-beneficiary of a social security system
* During a period of relative exclusion compared to another protocol
* Patient born before 36 weeks of amenorrhea
* Patient with a documented history of pulmonary fibrosis, primary pulmonary hypertension, cystic fibrosis, pulmonary malformation or chronic viral infections (hepatitis, HIV).
* Patient with any dental, nasopharyngeal or bronchial infection with fever (> 38°C) requiring systemic antibiotics in the previous 4 weeks

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2022-10-28 (Actual); Primary Completion 2025-04-28 (Estimated); Study Completion 2025-04-28 (Estimated)

PRIMARY OUTCOMES:
number of viral particles - Rhinovirus - Children -24 | after 24 hours of infection
  number of viral particles produced at the apical level after 24 hours of infection (Rhinovirus) by epithelia reconstituted in-vitro from samples from children
number of viral particles - Adenovirus - Children -24 | after 24 hours of infection
  number of viral particles produced at the apical level after 24 hours of infection (Adenovirus) by epithelia reconstituted in-vitro from samples from children
number of viral particles - SARS-CoV-2 - Children-24 | after 24 hours of infection
  number of viral particles produced at the apical level after 24 hours of infection (SARS-CoV-2 ) by epithelia reconstituted in-vitro from samples from children
number of viral particles - Rhinovirus - Adults-24 | after 24 hours of infection
  number of viral particles produced at the apical level after 24 hours of infection (Rhinovirus) by epithelia reconstituted in-vitro from samples from adults
number of viral particles - Adenovirus - Adults-24 | after 24 hours of infection
  number of viral particles produced at the apical level after 24 hours of infection (Adenovirus) by epithelia reconstituted in-vitro from samples from adults
number of viral particles - SARS-CoV-2 - Adults-24 | after 24 hours of infection
  number of viral particles produced at the apical level after 24 hours of infection (SARS-CoV-2 ) by epithelia reconstituted in-vitro from samples from adults
number of viral particles - Rhinovirus - elderly-24 | after 24 hours of infection
  number of viral particles produced at the apical level after 24 hours of infection ( Rhinovirus) by epithelia reconstituted in-vitro from samples from elderly people
number of viral particles - Adenovirus - Elderly-24 | after 24 hours of infection
  number of viral particles produced at the apical level after 24 hours of infection (Adenovirus) by epithelia reconstituted in-vitro from samples from elderly people.
number of viral particles - SARS-CoV-2 - Elderly-24 | after 24 hours of infection
  number of viral particles produced at the apical level after 24 hours of infection (SARS-CoV-2 ) by epithelia reconstituted in-vitro from samples from elderly people.

SECONDARY OUTCOMES:
number of viral particles - Rhinovirus - Children-48 | after 48 hours of infection
  number of viral particles produced at the apical level after 48 hours of infection (Rhinovirus) by epithelia reconstituted in-vitro from samples from children
number of viral particles - Rhinovirus - Children-72 | after 72 hours of infection
  number of viral particles produced at the apical level after 72 hours of infection (Rhinovirus) by epithelia reconstituted in-vitro from samples from children
number of viral particles - Rhinovirus - Children-96 | after 96 hours of infection
  number of viral particles produced at the apical level after 96 hours of infection (Rhinovirus) by epithelia reconstituted in-vitro from samples from children
number of viral particles - Rhinovirus - Children-168 | after 168 hours of infection
  number of viral particles produced at the apical level after 168 hours of infection (Rhinovirus) by epithelia reconstituted in-vitro from samples from children
number of viral particles - Adenovirus - Children -48 | after 48 hours of infection
  number of viral particles produced at the apical level after 48 hours of infection (Adenovirus) by epithelia reconstituted in-vitro from samples from children
number of viral particles - Adenovirus - Children -72 | after 72 hours of infection
  number of viral particles produced at the apical level after 72 hours of infection (Adenovirus) by epithelia reconstituted in-vitro from samples from children
number of viral particles - Adenovirus - Children -96 | after 96 hours of infection
  number of viral particles produced at the apical level after 96 hours of infection (Adenovirus) by epithelia reconstituted in-vitro from samples from children
number of viral particles - Adenovirus - Children -168 | after 168 hours of infection
  number of viral particles produced at the apical level after 168 hours of infection (Adenovirus) by epithelia reconstituted in-vitro from samples from children
number of viral particles - SARS-CoV-2 - Children-48 | after 48 hours of infection
  number of viral particles produced at the apical level after 48 hours of infection (SARS-CoV-2 ) by epithelia reconstituted in-vitro from samples from children
number of viral particles - SARS-CoV-2 - Children-72 | after 72 hours of infection
  number of viral particles produced at the apical level after 72 hours of infection (SARS-CoV-2 ) by epithelia reconstituted in-vitro from samples from children
number of viral particles - SARS-CoV-2 - Children-96 | after 96 hours of infection
  number of viral particles produced at the apical level after 96 hours of infection (SARS-CoV-2 ) by epithelia reconstituted in-vitro from samples from children
number of viral particles - SARS-CoV-2 - Children-168 | after 168 hours of infection
  number of viral particles produced at the apical level after 168 hours of infection (SARS-CoV-2 ) by epithelia reconstituted in-vitro from samples from children
number of viral particles - Adenovirus - Adults-48 | after 48 hours of infection
  number of viral particles produced at the apical level after 48 hours of infection (Adenovirus) by epithelia reconstituted in-vitro from samples from adults
number of viral particles - Adenovirus - Adults-72 | after 72 hours of infection
  number of viral particles produced at the apical level after 72 hours of infection (Adenovirus) by epithelia reconstituted in-vitro from samples from adults
number of viral particles - Adenovirus - Adults-96 | after 96 hours of infection
  number of viral particles produced at the apical level after 96 hours of infection (Adenovirus) by epithelia reconstituted in-vitro from samples from adults
number of viral particles - Adenovirus - Adults-168 | after 168 hours of infection
  number of viral particles produced at the apical level after 168 hours of infection (Adenovirus) by epithelia reconstituted in-vitro from samples from adults
number of viral particles - Rhinovirus - Adults-48 | after 48 hours of infection
  number of viral particles produced at the apical level after 48 hours of infection (Rhinovirus) by epithelia reconstituted in-vitro from samples from adults
number of viral particles - Rhinovirus - Adults-72 | after 72 hours of infection
  number of viral particles produced at the apical level after 72 hours of infection (Rhinovirus) by epithelia reconstituted in-vitro from samples from adults
number of viral particles - Rhinovirus - Adults-96 | after 96 hours of infection
  number of viral particles produced at the apical level after 96 hours of infection (Rhinovirus) by epithelia reconstituted in-vitro from samples from adults
number of viral particles - Rhinovirus - Adults-168 | after 168 hours of infection
  number of viral particles produced at the apical level after 168 hours of infection (Rhinovirus) by epithelia reconstituted in-vitro from samples from adults
number of viral particles - SARS-CoV-2 - Adults-48 | after 48 hours of infection
  number of viral particles produced at the apical level after 48 hours of infection (SARS-CoV-2 ) by epithelia reconstituted in-vitro from samples from adults
number of viral particles - SARS-CoV-2 - Adults-72 | after 72 hours of infection
  number of viral particles produced at the apical level after 72 hours of infection (SARS-CoV-2 ) by epithelia reconstituted in-vitro from samples from adults
number of viral particles - SARS-CoV-2 - Adults-96 | after 96 hours of infection
  number of viral particles produced at the apical level after 96 hours of infection (SARS-CoV-2 ) by epithelia reconstituted in-vitro from samples from adults
number of viral particles - SARS-CoV-2 - Adults-168 | after 168 hours of infection
  number of viral particles produced at the apical level after 168 hours of infection (SARS-CoV-2 ) by epithelia reconstituted in-vitro from samples from adults
number of viral particles - Rhinovirus - elderly-48 | after 48 hours of infection
  number of viral particles produced at the apical level after 48 hours of infection ( Rhinovirus) by epithelia reconstituted in-vitro from samples from elderly people
number of viral particles - Rhinovirus - elderly-72 | after 72 hours of infection
  number of viral particles produced at the apical level after 72 hours of infection ( Rhinovirus) by epithelia reconstituted in-vitro from samples from elderly people
number of viral particles - Rhinovirus - elderly-96 | after 96 hours of infection
  number of viral particles produced at the apical level after 96 hours of infection ( Rhinovirus) by epithelia reconstituted in-vitro from samples from elderly people
number of viral particles - Rhinovirus - elderly-168 | after 168 hours of infection
  number of viral particles produced at the apical level after 168 hours of infection ( Rhinovirus) by epithelia reconstituted in-vitro from samples from elderly people
number of viral particles - Adenovirus - Elderly-48 | after 48 hours of infection
  number of viral particles produced at the apical level after 48 hours of infection (Adenovirus) by epithelia reconstituted in-vitro from samples from elderly people.
number of viral particles - Adenovirus - Elderly-72 | after 72 hours of infection
  number of viral particles produced at the apical level after 72 hours of infection (Adenovirus) by epithelia reconstituted in-vitro from samples from elderly people.
number of viral particles - Adenovirus - Elderly-96 | after 96 hours of infection
  number of viral particles produced at the apical level after 96 hours of infection (Adenovirus) by epithelia reconstituted in-vitro from samples from elderly people.
number of viral particles - Adenovirus - Elderly-168 | after 168 hours of infection
  number of viral particles produced at the apical level after 168hours of infection (Adenovirus) by epithelia reconstituted in-vitro from samples from elderly people.
number of viral particles - SARS-CoV-2 - Elderly-48 | after 48 hours of infection
  number of viral particles produced at the apical level after 48 hours of infection (SARS-CoV-2 ) by epithelia reconstituted in-vitro from samples from elderly people.
number of viral particles - SARS-CoV-2 - Elderly-72 | after 72 hours of infection
  number of viral particles produced at the apical level after 72 hours of infection (SARS-CoV-2 ) by epithelia reconstituted in-vitro from samples from elderly people.
number of viral particles - SARS-CoV-2 - Elderly-96 | after 96 hours of infection
  number of viral particles produced at the apical level after 96 hours of infection (SARS-CoV-2 ) by epithelia reconstituted in-vitro from samples from elderly people.
number of viral particles - SARS-CoV-2 - Elderly-168 | after 168 hours of infection
  number of viral particles produced at the apical level after 168 hours of infection (SARS-CoV-2 ) by epithelia reconstituted in-vitro from samples from elderly people.

CONTACTS AND LOCATIONS:
Overall Officials: Michael FAYON, MDPhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No